CLINICAL TRIAL: NCT01772212
Title: Bioequivalence Study Between Two Medications for the Oral Administration of Terbinafine 250 mg in Oral Solids in Healthy Volunteers
Brief Title: Bioequivalence Study for Terbinafine 250 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 116827
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Mycoses
Keywords: Mexico; terbinafine; mycoses; pharmacokinetics
MeSH Terms: conditions — Mycoses | interventions — Terbinafine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A(test)/B(reference) (Experimental): Initial administration of test and crossover to reference
  Interventions: Drug: Terbinafine 250 mg
- B(reference)/A(test) (Experimental): Initial administration of reference and crossover to test
  Interventions: Drug: Terbinafine 250 mg

INTERVENTIONS:
Drug: Terbinafine 250 mg — Test product
  Other Names: Xilatril® is a registered trademark of Laboratorios Dermatológicos Darier
Drug: Terbinafine 250 mg — Reference product
  Other Names: Lamisil® is a registered trademark of Novartis

SUMMARY:
The objective of this study was to confirm if two formulations of terbinafine (tablets) are bioequivalent.

Test product was Xilatril® 250 mg (Laboratorios Dermatológicos Darier) and reference product Lamisil® 250 mg (Novartis). One tablet was the single dosage.

The study was prospective, open-label, randomized, crossover, single dose, with 02 treatments, 02 sequences and 02 periods, under fasting conditions.

The population was composed of 30 healthy volunteers, both genders, adults between 18-50 years.

The comparative bioavailability of the two formulations was evaluated based in statistical comparisons of relevant pharmacokinetic parameters, obtained from data of drug concentrations in blood.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria: Males 18-50 years. Healthy based on comprehensive medical history, lab tests, Chest x-ray, Electrocardiogram, negative tests for Hepatitis B and C, and HIV. Negative urine doping test. BMI 19-26.5 kg/m2. Lab test in normal range +/- 10%. Blood pressure 139-90/89-50, heart rate 100-55, respiratory rate 24-17, temperature 37.5-35 °C. Non-smoking at least for 10 hrs before study. Written informed consent. -

Exclusion Criteria:

Hypersensitivity to study medication or other related drug. History of cardiovascular, renal, hepatic, metabolic, gastrointestinal, neurologic, endocrine, hematopoietic, psychiatric or organic condition.

Requiring any drug interfering with minocycline pharmacokinetics. Exposed to inducers or inhibitors of hepatic enzymes. Intake of possible toxic drugs 30 days before study. Intake of any drug 14 days or 7 half-lives before study. Hospitalization or severe disease 60 days before study. Receiving investigational drug out of study center 30 days before study. Blood loss or blood donation =>450 ml 60 days before study. Recent history of drug abuse including alcohol. Intake of xanthine containing products 10 hrs before study. Intake of grapefruit juice or hot-spice 10 hrs before study.

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02-24 (Actual); Primary Completion 2011-03-15 (Actual); Study Completion 2011-03-15 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (CMAX) of drug terbinafine | 0.0, 0.33, 0.66, 1.0, 1.33, 1.66, 2.0, 2.33, 2.66, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, and 24.0 hours post dose
  pharmacokinetics
Area under the plasma concentration versus time curve (AUC) of drug terbinafine | 0.0, 0.33, 0.66, 1.0, 1.33, 1.66, 2.0, 2.33, 2.66, 3.0, 3.5, 4.0, 6.0, 8.0, 10.0, 12.0, and 24.0 hours post dose
  pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- See also: Results for study 116827 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116827?search=study&search_terms=116827#rs